CLINICAL TRIAL: NCT01982097
Title: Multicenter, Prospective, Non-interventional Study "Sorafenib as Neoadjuvant Therapy Before Cytoreductive Nephrectomy in Patients With Metastatic Renal Cell Carcinoma"
Brief Title: Sorafenib as Neoadjuvant Therapy Before Cytoreductive Nephrectomy in Patients With Metastatic Renal Cell Carcinoma
Acronym: SANE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16933; NX1307RU (Other: company internal)
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Carcinoma, Renal Cell
Keywords: Non-interventional; Nexavar; Sorafenib; Carcinoma, renal cell; Neoadjuvant; Nephrectomy; Russian Federation
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY 43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY 43-9006) — The patients under routine treatment of metastatic RCC with Nexavar before and after cytoreductive nephrectomy meeting the criteria of inclusion.

SUMMARY:
This local, prospective, multicenter, non-interventional study documents observational data on patients under routine treatment of metastatic RCC with Nexavar before and after cytoreductive nephrectomy. It's planned to better understand the impact of cytoreductive nephrectomy on Nexavar efficacy and possibly to define patients who get the most benefit from Nexavar before cytoreductive nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* - Male and female patients ≥ 18 years old
* Patients with untreated metastatic RCC in whom a decision on neoadjuvant treatment with Nexavar before cytoreductive nephrectomy and in case of clinical feasibility resumption of treatment with Nexavar after nephrectomy has been made at the time of study enrollment
* Life expectancy of at least 16 weeks
* Patients should have signed informed consent form

Exclusion Criteria:

* Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell carcinoma, squamous cell skin cancer, or in situ cervical cancer.
* All contra-indications according to the Russian marketing authorization:

  * Hypersensitivity to sorafenib or to any of the excipients.
  * Pregnancy and breast-feeding.
  * Age less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients ≥ 18 years old with untreated metastatic RCC for whom treatment with Nexavar is planned with subsequent cytoreductive nephrectomy and resumption of Nexavar in case of clinical feasibility
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Maximum percent reduction (based on the minimum post baseline value) in the longest diameter of the primary tumor in response to neoadjuvant Nexavar treatment. | up to 2 years
Response rate of residual disease to Nexavar according to RECIST 1.1 with baseline after cytoreductive nephrectomy. | up to 2 years

SECONDARY OUTCOMES:
Response before cytoreductive nephrectomy according to RECIST 1.1. | up to 2 years
Maximum percent reduction in the sum of longest diameters of target lesions according to RECIST 1.1 while on Nexavar treatment before cytoreductive nephrectomy | up to 2 years
Maximum percent reduction in the sum of longest diameters of target lesions of residual disease after cytoreductive nephrectomy according to RECIST 1.1 while on Nexavar treatment with baseline after cytoreductive nephrectomy. | up to 2 years
Number of participants with AEs, including intra- and postoperative complications, relation to Nexavar treatment, AEs treatment, AEs outcome. | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Russia